CLINICAL TRIAL: NCT02880683
Title: Cardiac Output Autonomic Stimulation Therapy for Heart Failure (COAST-HF) - Human NeuroCatheter Study
Acronym: COAST-HF HNrCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroTronik Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 700019-01
Record Dates: First submitted 2016-08-10; First posted 2016-08-26 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Output, Low
Keywords: Electrical Stimulation Therapy; Parasympathetic Nervous System; Sympathetic Fibers; Post Ganglionic; Congestive Heart Failure; Heart Failure
MeSH Terms: conditions — Cardiac Output, Low; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm, transvenous cardiac autonomic nerve stimulation (Experimental)
  Interventions: Device: NeuroTronik CANS Therapy System

INTERVENTIONS:
Device: NeuroTronik CANS Therapy System

SUMMARY:
A single-center feasibility study in patients undergoing cardiac catheterization, to investigate the acute hemodynamic effects of transvenous cardiac autonomic nerve stimulation.

DETAILED DESCRIPTION:
A single-center feasibility study performed in patients undergoing a planned cardiac catheterization. This study investigated the feasibility of the NeuroTronik CANS Therapy™ System to improve acute hemodynamics. Purpose-built stimulation catheters were percutaneously inserted into an upper venous structure near the heart via right femoral vein and or left subclavian vein access using standard introducers and techniques. Subjects were instrumented with left ventricular and femoral artery catheters for pressure measurement and stimulated for approximately 60 minutes. Baseline hemodynamic measures were collected before stimulation and compared to measured values during stimulation. Following completion of the protocol, all in-dwelling equipment and catheters were removed.

ELIGIBILITY:
Inclusion Criteria:

* Stable symptomatic heart failure - New York Heart Association Class II or III
* Normal Sinus Rhythm

Exclusion Criteria:

* Unable to gain arterial or venous access using standard percutaneous techniques
* New York Heart Association Class IV
* Patient taking amiodarone or other anti-arrhythmic therapy
* Patients with implanted pacemaker, ICD, or CRT device
* Patients who had CABG, PCI or enzyme-positive MI within prior month
* Patients with pre-existing carotid artery or cerebral disease
* Patients with hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis)
* Patients who have been hospitalized for heart failure and who required the use of heart failure IV therapy within 30 days before enrollment (measured from release)
* Patients with current or prior vagal nerve simulator
* Patients with renal failure
* Patients with hepatic failure
* Patients with narrow angle glaucoma
* Patients who are pregnant
* Patients with a life expectancy < 12 months per physician judgment
* Patients with allergy to fentanyl, midazolam, propofol, eggs, egg products, soybeans, or soy products

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cardiac output | One hour

SECONDARY OUTCOMES:
Arterial blood pressure | One hour
Left ventricular pressure | One hour
Heart rate | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, Medical Doctor, Principal Investigator — Facultad de Ciencias Medicas UNA Paraguay, Asuncion, Paraguay
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided